CLINICAL TRIAL: NCT01664975
Title: A Randomized Controlled Multi-center Clinical Trial on Treatment of Peripheral T-cell Lymphoma With DGPT Regiment (Gemcitabine,Cisplatin,Prednisone ,Thalidomide )
Brief Title: Treatment of Peripheral T-cell Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mingzhi Zhang (Other)
Collaborators: Zhengzhou University (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx2011-3
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-08

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: Peripheral T-cell lymphoma;chemotherapy;; RR;PFS;OS
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — VAP-cyclo protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GDPT regimen (Experimental): GDPT(gemcitabine,cisplatin,Prednisone,Thalidomide) regimen
  Interventions: Drug: GDPT regimen
- CHOP regimen (Experimental): CHOP(Cyclophosphamide,Vincristine,Doxorubicin,Prednisone) regimen
  Interventions: Drug: CHOP regimen

INTERVENTIONS:
Drug: GDPT regimen — GDPT regimen(Gemcitabine,Cisplatin,Prednisone ,Thalidomide) Cisplatin(DDP) 25 mg/m2,ivgtt（intravenously guttae）,d1-3;Prednisone 60mg/m2,p.o,d1-5;Gemcitabine(GEM) 800mg/m2,ivgtt,30min,d1,8;Thalidomide,p.o,200mg/d,Continued use to the end of chemotherapy .Every 21 days for one cycle and three cycles are required. Efficacy was evaluated every two cycles.
  Arms: GDPT regimen
Drug: CHOP regimen — CHOP regimen(Cyclophosphamide,Vincristine,Doxorubicin,Prednisone) Cyclophosphamide 750mg/d,ivgtt, d1;Vincristine,1.4g/m2,ivgtt, d1;Doxorubicin,50mg/m2,ivgtt,d1;Prednisone 60mg/m2,p.o, d1-5.
  Arms: CHOP regimen

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of GDPT regiment (gemcitabine，cisplatin,Prednisone ,Thalidomide

) for patients with Peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
Patients with Peripheral T-cell lymphoma usually have a bad prognosis. These patients cannot be treated successfully with the conventional chemotherapy of CHOP. The investigators have been proceeding this trial to evaluate the efficacy and safety of the combination chemotherapy regiment GDPT regiment (gemcitabine，cisplatin,Prednisone ,Thalidomide

) in the patients with Peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Age range 14-70 years old; ECOG performance status 0-2; Estimated survival time > 3 months Histological confirmed Peripheral T cell lymphoma None of chemotherapy or radiotherapy has been previously used None of chemotherapy contraindication: hemoglobin ≥ 90 g/dl, neutrophil ≥ 1.5×109/L, platelet ≥ 100×109/L, ALT and AST ≤ 2×ULN, serum bilirubin ≤ 1.5×ULN, serum creatine ≤ 1.5×upper limitation of normal (ULN), Serum Albumin ≥ 30g/L, serum plasminogen is normal (Inclusion Criteria of 1,3,6 groups ) At least one measurable lesion None of other serious diseases, cardiopulmonary function is normal Pregnancy test of women at reproductive age must be negative Patients could be followed up None of other relative treatments including the traditional Chinese medicine, immunotherapy,biotherapy except anti-bone metastasis therapy and other symptomatic treatments.

volunteers who signed informed consent.

Exclusion Criteria:

Disagreement on blood sample collection Patients allergic of any of drug in this regimen or with metabolic disorder Pregnant or lactating women Serious medical illness likely to interfere with participation Serious infection Primitive or secondary tumors of central nervous system Chemotherapy or radiotherapy contraindication The evidence of CNS metastasis History of peripheral nervous disorder or dysphrenia patients participating in other clinical trials patients taking other antitumor drugs patients estimated to be unsuitable by investigato

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi Zhang, Pro,Dr, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Sun Y, Li L, Li X, Zhang L, Wang X, Fu X, Sun Z, Zhang X, Li Z, Wu J, Yu H, Chang Y, Yan J, Wu X, Zhou Z, Nan F, Tian L, Zhang M. Outcomes of GDPT (gemcitabine, cisplatin, prednisone, thalidomide) versus CHOP in newly diagnosed peripheral T-cell lymphoma patients. Ther Adv Med Oncol. 2020 May 27;12:1758835920923829. doi: 10.1177/1758835920923829. eCollection 2020. PMID 32550864
- [Derived] Li L, Duan W, Zhang L, Li X, Fu X, Wang X, Wu J, Sun Z, Zhang X, Chang Y, Nan F, Yan J, Li Z, Young KH, Zhang M. The efficacy and safety of gemcitabine, cisplatin, prednisone, thalidomide versus CHOP in patients with newly diagnosed peripheral T-cell lymphoma with analysis of biomarkers. Br J Haematol. 2017 Sep;178(5):772-780. doi: 10.1111/bjh.14763. Epub 2017 Jun 9. PMID 28597542

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GDPT Regimen | CHOP Regimen
Started | 57 | 54
Completed | 52 | 51
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GDPT Regimen | CHOP Regimen | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 43 | 46 | 89
  >=65 years | 8 | 4 | 12
Age, Continuous [Median (Full Range); unit: years] | 55 [16 to 69] | 51 [15 to 70] | 55 [15 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 31 | 47
  Male | 36 | 20 | 56
Region of Enrollment [Number; unit: participants]
  China | 52 | 51 | 103

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Time Frame: up to end of follow-up-phase (approximately 24 months)
Measure: Number; unit: participants
Arm/Group | GDPT Regimen | CHOP Regimen
Number analyzed (Participants) | 52 | 51
participants | 35 | 27

2. Secondary Outcome: Response Rate
Description: 21 days(3 weeks) for one cycle,Efficacy was evaluated every two cycles
Time Frame: every 6 weeks,up to completion of treatment(approximately 18 weeks )
Reporting Status: Not Posted, anticipated posting 2016-09

3. Secondary Outcome: Overall Survival
Time Frame: up to the date of death (approximately 5 years)
Reporting Status: Not Posted, anticipated posting 2016-09

4. Secondary Outcome: Median Survival Time
Time Frame: 24 months
Reporting Status: Not Posted, anticipated posting 2016-12

ADVERSE EVENTS:
Arm/Group | GDPT Regimen | CHOP Regimen
Serious Adverse Events (participants affected / at risk) | 23/52 | 21/51
Other Adverse Events (participants affected / at risk) | 21/52 | 19/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GDPT Regimen (N=52) | CHOP Regimen (N=51)
Grade3/4 myelosuppression (Blood and lymphatic system disorders) | 23 | 21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GDPT Regimen (N=52) | CHOP Regimen (N=51)
digestive tract toxicity (Gastrointestinal disorders) | 21 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes